CLINICAL TRIAL: NCT01262833
Title: A Cohort Study of the Functional Significance of Internal Pudendal Artery Stenoses in Patients With Erectile Dysfunction
Brief Title: Pudendal Assessment in Erectile Dysfunction
Acronym: INDEED
Status: Terminated | Type: Observational
Why Stopped: data suggesting pudendal artery stenosis rarely being cause of ED
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Other Study IDs: 811936
Record Dates: First submitted 2010-11-12; First posted 2010-12-17 (Estimated); Last update posted 2014-03-14 (Estimated); Status verified 2012-01

CONDITIONS: Erectile Dysfunction
MeSH Terms: conditions — Erectile Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Cases: Patients with erectile dysfunction by ILEF questionnaire
- Controls: Patients without erectile dysfunction by ILEF questionnaire

SUMMARY:
The study will address the role of internal pudendal artery disease in erectile dysfunction (ED), and whether it might eventually be amenable to intervention with stenting. There is currently a small trial investigating the potential benefit of stenting for erectile dysfunction, but the relationship between pelvic arterial stenoses and erectile dysfunction is not yet proven. The investigators intend to perform angiography on patients both with and without erectile dysfunction, to see whether internal pudendal artery disease is more common in the population with erectile dysfunction. In addition to angiography, stenoses will be examined using fractional flow reserve. The degree of internal pudendal artery disease will then be correlated with the degree of erectile dysfunction using a validated questionnaire, the International Index of Erectile Function (IIEF). Patients will then complete IIEF questionnaires for 5 years to assess the relationship between internal pudendal artery disease and progression of erectile dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* As above, men with one risk factor for ED such as age>55, diabetes, hyperlipidemia, smoking, hypertension, coronary disease or peripheral arterial disease

Exclusion Criteria:

* Patients with ED from a non-arterial cause, including hormonal, neurological, or trauma-related (as determined by past medical history routinely performed prior to catheterization)
* Patients requiring urgent catheterization (e.g. acute coronary syndrome or cardiogenic shock)
* Patients with a creatinine >1.5 mg/dL and those deemed at increased renal risk (such as from receiving >200 mL of dye during the primary procedure, post renal transplant or single kidney), as the additional contrast dye required for angiography would pose an undue risk of progressive kidney disease
* Patients with other illnesses that reduce their life expectancy to less than one year

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: sexually active men, scheduled for cardiac catheterization or peripheral artery catheterization, who have at least one risk factor for ED
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2010-09; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Pudendal Assessment in Erectile Dysfunction | Up to Five years
  The primary exposure will be hemodynamically significant internal pudendal artery stenoses as a predictor of erectile dysfunction

SECONDARY OUTCOMES:
Pudendal Assessment in Erectile Dysfunction | up to five years
  Secondary analyses will include correlation between bilateral disease and erectile dysfunction, as well as the contribution of small vessel disease (distal to the internal pudendal artery). The severity of disease by IIEF questionnaire will also be compared to the severity of disease by angiography. We will continue through 5-year follow-up of patients with yearly IIEF questionnaires to determine if changes in erectile dysfunction can be predicted by baseline internal pudendal artery disease.

CONTACTS AND LOCATIONS:
Overall Officials: Howard Herrmann, M.D., Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States